CLINICAL TRIAL: NCT00759525
Title: The Role of Mineralocorticoid Receptors in Vascular Function
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Joshua A. Beckman, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2001-P-001404
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Results first posted 2015-05-28 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-09

CONDITIONS: Apparent Mineralocorticoid Excess (AME)
MeSH Terms: conditions — Mineralocorticoid Excess Syndrome, Apparent | interventions — Glycyrrhetinic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Glycyrrhetic Acid
  Interventions: Drug: Glycyrrhetic Acid
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Glycyrrhetic Acid — 130 mg daily for fourteen days
  Other Names: licorice root sweetener
  Arms: 1
Drug: Placebo — Placebo daily for fourteen days
  Arms: 2

SUMMARY:
The purpose of this study is to figure out how decreasing the activity of 11-beta hydroxysteroid dehydrogenase (11-beta HSD) will affect your blood vessel function. 11-beta HSD, which is found in the kidneys and blood vessels, is a natural protein that when active helps to keep your blood pressure under control.

DETAILED DESCRIPTION:
This study intends to determine whether activation of mineralocorticoid receptors affects vascular function. Vascular function relies on two components of the blood vessel: the inner lining (endothelium) and the vascular smooth muscle. In specific aim 1, we seek to determine if that inhibition of the enzyme 11-beta hydroxysteroid dehydrogenase (11-beta-HSD) will impair endothelium-dependent vasodilation and/or vascular smooth muscle function.

The syndrome of apparent mineralocorticoid excess (AME) is a rare disorder identified in approximately 50 individuals characterized by low-aldosterone hypertension, associated with low renin and hypokalemia These subjects avidly retain salt and water, have suppression of both plasma renin and aldosterone levels, but clinically appear as though they have a state of mineralocorticoid excess. A detailed series of investigations has elucidated the cause of this syndrome: severe attenuation of the enzyme 11 beta-hydroxysteroid dehydrogenase (11-beta-HSD). 11-beta-HSD converts cortisol, able to activate mineralocorticoid receptors to cortisone, which cannot. This abnormality can be identified by measuring an abnormal ratio of urinary breakdown products of cortisol and cortisone. Subjects with AME have a high ratio indicative of elevated cortisol concentrations.

Although classical AME is a rare syndrome with a specific recessive inheritance, several other mutations have been identified which cause a varying severity of disease. Recent evidence has suggested mild abnormalities in this pathway may be much more common. In fact two studies have demonstrated that subjects with essential hypertension had greater levels of cortisol/cortisone urinary levels than matched controls. Thus, mild abnormalities of this enzyme may be an important contributor to a segment of patients with high blood pressure. Further, this is the pathway by which consumption of excess black licorice causes hypertension. Black licorice contains glycyrrhizic acid that selectively inhibits 11 beta-HSD. Glycyrrhizic acid is used as a dietary sweetener and sold in "health-food" stores and may also play a epidemiological role in hypertension.

Analogous to the renin-angiotensin system, 11-beta-HSD is not only found in the kidneys, but is found in both vascular endothelial (inner lining) and smooth muscle cells. Hypertension, similar to other risk factors for cardiovascular disease impairs vascular function. One of its major effects is decreasing the bioavailability of endothelium-derived nitric oxide. Nitric oxide contributes importantly to vascular homeostasis by modulating vascular tone, inhibiting both platelet aggregation and coagulation, and inhibition translocation of leukocytes into the vascular wall. Further, patients with hypertension have increased endothelin-1 production and receptor activation. Endothelin-1 antagonizes the beneficial activities of nitric oxide. Experimentally, inactivation of 11 beta-HSD in a rat model has been demonstrated to cause hypertension, increase endothelin receptor A activation and decrease bioavailability of endothelium-derived nitric oxide. Inhibition of mineralocorticoid receptors in this model prevents impairment of vascular function. Thus, in animal models, abnormalities in this pathway may not only cause hypertension, but create an environment favorable to the development and progression of atherosclerosis. Further, recent evidence suggests that activation of this pathway contributes importantly to the morbidity and mortality in patients with congestive heart failure. A large, randomized study demonstrated that a small dose of a mineralocorticoid inhibitor, spironolactone, substantially reduced morbidity and mortality in patients with severe heart failure. Experimentally, spironolactone improved vascular function in patients with congestive heart failure.

Therefore, we seek to characterize the vascular effects of this pathway in humans. This submission involves one protocol: 1) to determine if reversible inhibition of 11 beta-HSD decreases the bioavailability of endothelium-derived nitric oxide and impairs vascular smooth muscle function.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Blood pressure above 140/90
* Abnormal physical finding
* Blood test values for total and LDL cholesterol, CBC, sodium, potassium, creatinine, and glucose laboratories greater 1.5 times normal

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2002-02; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua A Beckman, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Sobieszczyk P, Borlaug BA, Gornik HL, Knauft WD, Beckman JA. Glycyrrhetinic acid attenuates vascular smooth muscle vasodilatory function in healthy humans. Clin Sci (Lond). 2010 Aug 5;119(10):437-42. doi: 10.1042/CS20100087. PMID 20515440
- See also: Glycyrrhetinic acid attenuates vascular smooth muscle vasodilatory function in healthy humans. — http://www.ncbi.nlm.nih.gov/pubmed/?term=Joshua+Beckman+mineralocorticoid

RESULTS

PARTICIPANT FLOW:
Groups:
- Glycyrrhetinic Acid First, Then Placebo: Glycyrrhetic Acid-130 mg/day for 14 days followed by placebo
- Placebo First, Then Glycyrrhetinic Acid: Placebo followed by Glycyrrhetic Acid-130 mg/day for 14 days
Period: First Intervention (14 Days)
Arm/Group | Glycyrrhetinic Acid First, Then Placebo | Placebo First, Then Glycyrrhetinic Acid
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0
Period: Washout (14 Days)
Arm/Group | Glycyrrhetinic Acid First, Then Placebo | Placebo First, Then Glycyrrhetinic Acid
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0
Period: Second Intervention (14 Days)
Arm/Group | Glycyrrhetinic Acid First, Then Placebo | Placebo First, Then Glycyrrhetinic Acid
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Cross Over study
Arm/Group | All Study Participants
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Forearm Blood Flow
Description: At the end of each 14-day intervention (Glycyrrhinitic acid or Placebo), vascular endothelial function was assessed by measuring forearm blood flow and comparing to Baseline. The outcome measure depicted below reflects the change in forearm blood flow from Baseline after completing the glycyrrhinitic acid regimen as well as the change in forearm blood flow from Baseline after taking the matching placebo.
Time Frame: Outcome was measured at the end of each study period (i.e. 14 days after Baseline measurements were taken)
Measure: Mean (Standard Error); unit: ml/100ml of tissue/min
Groups:
- Glycyrrhinitic Acid; Placebo: All of the 15 subjects received both glycyrrhinitic acid (130mg/day) (GA) for a 14-day period and placebo for a 14-day period. Approximately half of the subjects received GA before placebo; the other half received placebo before GA. There was a 2-week washout period between the two conditions.
Arm/Group | Glycyrrhinitic Acid | Placebo
Number analyzed (Participants) | 15 | 15
ml/100ml of tissue/min | 1.87 (0.26) | 1.34 (0.20)

ADVERSE EVENTS:
Time Frame: 30 days.
Description: Subjects were queried concerning their catheter insertion site.
Groups:
- Glycyrrhetinic Acid First, Then Placebo; Placebo First, Then Glycyrrhetinic Acid: Healthy subjects without medical condition.
Arm/Group | Glycyrrhetinic Acid First, Then Placebo | Placebo First, Then Glycyrrhetinic Acid
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No